CLINICAL TRIAL: NCT06021483
Title: Observational Study to Evaluate the Safety and Efficacy of Zepzelca™ Injection (Lurbinectedin) in Patients With Metastatic Small Cell Lung Cancer (SCLC) in Real-World Practice
Brief Title: Observational Study to Evaluate the Safety and Efficacy of Zepzelca™ Injection
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-LTD-OS-401
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: SCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Zepzelca™ inj. in real-world practice and to investigate important identified risks and gaps in information related to risk management plans.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily provide written consent for personal information collection and utilization after receiving an explanation about the objective and methods of the study
* Patients who have received or are scheduled to receive Zepzelca™ inj., according to domestic approval indications
* Patients with metastatic SCLC who have failed first-line platinum-based chemotherapy

Exclusion Criteria:

* Patients with no prior history of platinum-based anticancer chemotherapy for cancer treatment
* Patients with a history of hypersensitivity reactions to this drug or its components
* Pregnant, potentially pregnant, or lactating women
* Patients currently participating in another clinical trial (drug or medical device) or planning to participate in another clinical trial during the study period (except for non-interventional clinical studies or cases where the clinical trial drug administration has ended and only follow-up is remaining)
* Patients who are judged by the principle Investigator or sub-Investigator to be ineligible to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Metastatic SCLC who have failed first-line platinum-based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
ORR (Overall Response Rate) | 6 months after the start of administration
  Percentage of subjects who reached complete remission (CR) and partial remission (PR)

OTHER OUTCOMES:
SAE & SADR Incidence Rate | 6 months after the start of administration
  Serious Adverse Event & Serious Adverse Drug Reaction Incidence Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Boramae Medical Center, Seoul, South Korea